CLINICAL TRIAL: NCT05593783
Title: The Use of the "Comprehensive Complication Index" as a Recording System of Postoperative Complications After Percutaneous, Retrograde and Extracorporeal Lithotripsy for Renal Lithiasis.
Brief Title: The Use of the "Comprehensive Complication Index" for Urinary Lithiasis Surgery.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sismanoglio General Hospital (Other)
Responsible Party: Principal Investigator, Stamatios Katsimperis, Dr Stamatios Katsimperis, Sismanoglio General Hospital
Other Study IDs: 67127
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Complication,Postoperative; Lithiasis, Urinary
Keywords: clavien dindo; urinary lithiasis; endourology; complications
MeSH Terms: conditions — Postoperative Complications; Urolithiasis | interventions — Lithotripsy; Nephrolithotomy, Percutaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with lithiasis treated with ureterolithotripsy: patients with lithiasis treated with ureterolithotripsy
  Interventions: Procedure: lithotripsy
- patients with lithiasis treated with percutaneous nephrolithotomy: patients with lithiasis treated with percutaneous nephrolithotomy
  Interventions: Procedure: lithotripsy
- patients with lithiasis treated with extracorporeal shockwave lithotripsy: patients with lithiasis treated with extracorporeal shockwave lithotripsy
  Interventions: Procedure: lithotripsy

INTERVENTIONS:
Procedure: lithotripsy — lithotripsy
  Other Names: percutaneous nephrolithotomy; extracorporeal shockwave lithotripsy

SUMMARY:
The study will be prospective non-interventional and will include patients with kidney stones who are to undergo one of the following three techniques: retrograde nephrolithotripsy, percutaneous nephrolithotripsy and extracorporeal nephrolithotripsy depending on the size of the stone. Data regarding post operative descriptions will be recorded and comprehensive complication index will be used for the assesment of the burden.

DETAILED DESCRIPTION:
The study will be prospective non-interventional and will include patients with kidney stones who are to undergo one of the following three techniques: retrograde nephrolithotripsy, percutaneous nephrolithotripsy and extracorporeal nephrolithotripsy depending on the size of the stone. The study will take place at the 2nd Urology Clinic of the University of Athens, at the Sismanoglio Hospital of Athens. It will include patients diagnosed with kidney stones after plain X-ray and/or CT scan. Percutaneous nephrolithotripsy will be performed on stones > 2 cm, while extracorporeal or retrograde nephrolithotripsy on stones < 2 cm. Patient demographics (age, gender, body mass index, comorbidities, anticoagulant use), stone-related data (maximum stone size, anatomic location of stone, number of stones, presence of hydronephrosis preoperatively, presence of piglet catheter preoperatively, positive urine culture, preoperative chemoprophylaxis ) as well as information about the operation (type of anesthesia, operation time, hospitalization time) will be reported. Finally, all possible complications will be recorded intraoperatively, immediately postoperatively and up to 30 days after the day of surgery. This will be followed by a statistical analysis of the resulting data and a comparison between the CDC and CCI systems using the SPSS statistical program. To describe continuous variables, the mean/standard deviation will be used if it is a normal distribution, or the median and range if it is a non-normal distribution. The Shapiro-Wilk test will be used to investigate the distribution of the data. The absolute number and the corresponding percentage will be used to describe the qualitative variables. For the comparison of continuous variables, the parametric t-test will be used if the data follow a normal distribution, or the Mann-Whitney U test if they do not follow a normal distribution. Chi-square and Fisher's exact test will be used to compare qualitative variables. Exclusion criteria from this study are:

1. Non-acceptance by the patient of his participation or inability to understand the purposes and procedures of the study.
2. Recent similar operation that the patient has undergone (interval of less than one month).

ELIGIBILITY:
Inclusion Criteria:

Patients with urinary lithiasis undergoing ureterolithotripsy, percutaneous nephrolithotripsy or extracorporeal shockwave lithotripsy.

Exclusion Criteria:

- 1. Non-acceptance by the patient of his participation or inability to understand the purposes and procedures of the study.

2. Recent similar operation that the patient has undergone (interval of less than one month).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with lithiasis
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
comprehensive complication index score | 1,5 year
  reporting postoperative complications with clavien dindo and comprehensive complication index and comparison of those two.

CONTACTS AND LOCATIONS:
Locations (1):
- Sismanoglio General Hospital, Athens, Marousi, Greece

IPD SHARING:
Plan to Share IPD: No